CLINICAL TRIAL: NCT00106899
Title: Alzheimer's Disease Neuroimaging Initiative
Brief Title: ADNI: Alzheimer's Disease Neuroimaging Initiative
Status: Completed | Type: Observational
Sponsor: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Collaborators: Northern California Institute of Research and Education (Other); National Institute on Aging (NIA) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Foundation for the National Institutes of Health (Other); Alzheimer's Drug Discovery Foundation (Other); Alzheimer's Association (Other)
Responsible Party: Sponsor
Other Study IDs: IA0068; 1RC2AG036535 (NIH); 1U01AG024904 (NIH)
Record Dates: First submitted 2005-03-31; First posted 2005-04-01 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Alzheimer's Disease
Keywords: neuroimaging; brain metabolism; biomarkers; cognition disorder; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognition Disorders; Cognitive Dysfunction | interventions — Magnetic Resonance Spectroscopy; Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Mild Cognitive Impairment (MCI); scans performed at screening/baseline, 6, 12, 18, 24, and 36 months
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Procedure: Positron Emission Tomography (PET); Procedure: Lumbar Puncture (LP)
- 2: Early Alzheimer's disease (AD); scans performed at screening/baseline, 6, 12, and 24 months
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Procedure: Positron Emission Tomography (PET); Procedure: Lumbar Puncture (LP)
- 3: Unaffected/normal controls; scans performed at baseline/screening, 6, 12, 24, and 36 months
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Procedure: Positron Emission Tomography (PET); Procedure: Lumbar Puncture (LP)

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — MRI scans
Procedure: Positron Emission Tomography (PET) — PET scans
Procedure: Lumbar Puncture (LP) — collection of cerebrospinal fluid
  Other Names: spinal tap

SUMMARY:
The purpose of this study is to examine how brain imaging technology can be used with other tests to measure the progression of mild cognitive impairment (MCI) and early Alzheimer's disease (AD). This information will aid future clinical trials by providing a standard assessment tool to measure the effects of treatments being studied.

DETAILED DESCRIPTION:
This study will test whether serial magnetic resonance imaging (MRI), positron emission tomography (PET), other biological markers, and clinical and neuropsychological assessment can be combined to measure the progression of mild cognitive impairment (MCI) and early Alzheimer's disease (AD). The information obtained by studying changes in the brain images of MCI and AD patients and healthy individuals, as well as other assessment tools, will be used to determine the best methods for measuring treatment effects in patients with MCI and AD.

Approximately 800 participants, ranging in age from 55 to 90, will be recruited for the study: 400 patients with MCI, 200 with early AD, and 200 normal controls. Patients with MCI and normal controls will be followed for 3 years, and those with AD will be followed for 2 years. At 6-month intervals, all participants will be seen in person or contacted by telephone. All participants will undergo repeated scanning and blood and urine biomarkers will be collected at the time of each scan. All patients will be asked if they are willing to undergo lumbar puncture at baseline and year one, with the goal of a minimum of 20% and as many as 50% of each group providing CSF (cerebrospinal fluid) samples for analysis and storage for future analyses.

NOTE: Beginning in Spring 2007 a subset of the ADNI participants will be offered the opportunity to participate in a supplemental study. The PIB (Pittsburgh Compound B) study provides imaging of amyloid plaque burden. PIB PET scans will be conducted in 24 control, 48 MCI, and 24 AD participants at approximately 16 ADNI PET sites. For entering participants with no previous PET FDG scans, controls and MCI participants will be scanned with PIB at entry (baseline), 12, 24, and 36 months, and AD participants will be scanned with PIB at entry (baseline), 12, and 24 months. For participants who have undergone previous (baseline and 6 month) PET FDG scans, controls and MCI participants will be scanned with PIB at 12, 24, and 36 months, and AD participants will be scanned with PIB at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

Participants will be classified as either MCI patients, AD patients, or normal controls. General Inclusion Criteria will apply to all groups, with specific criteria for each group as described below:

General (applies to each category):

* Between 55 and 90 years of age (Currently, ADNI sites are only recruiting volunteers age 70-90 among people with no memory problems)
* Study partner or caregiver to accompany patient to all scheduled visits
* Fluent in English or Spanish
* Permitted medications stable for at least 4 weeks prior to screening
* Adequate visual and auditory acuity to allow neuropsychological testing
* Good general health with no additional diseases expected to interfere with the study
* Women must be two years post-menopausal or surgically sterile
* Willing and able to complete all baseline assessments, and to participate in the 2-3 year protocol
* Willing to undergo neuroimaging and provide DNA and plasma samples as specified
* Completed 6 grades of education or sufficient work history to exclude mental retardation
* Modified Hachinski score <=4
* Geriatric Depression Scale <6

Specific Criteria for MCI and AD patients:

* Memory complaint by patient or study partner
* Abnormal memory function score on Wechsler Memory Scale (adjusted for education)
* Mini-Mental State Exam score between 24 and 30 (MCI) or 20 and 26 (AD)
* Clinical Dementia Rating = 0.5; Memory Box score at least 0.5 (MCI) or 1.0 (AD)

Exclusion Criteria:

* Any significant neurologic disease other than Alzheimer's disease
* Abnormal baseline MRI
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin, or body
* Major depression, bipolar disorder, history of schizophrenia
* History of alcohol or substance abuse or dependency within the past 2 years
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol
* Clinically significant laboratory abnormalities
* Residence in skilled nursing facility
* Participation in clinical studies involving neuropsychological measures being collected more than one time per year

Specific Exclusion Criteria for MCI and AD:

* Psychotic features, agitation or behavioral problems within the last 3 months which could lead to difficulty complying with the protocol.

Prohibited medications:

* Specific psychoactive medications (for example, certain antidepressants, anti-anxiety medications, sleeping pills, etc.)
* Warfarin (Coumadin)
* Investigational agents

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 818 (Actual)
Dates: Start 2005-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Weiner, MD, Principal Investigator — University of California, San Francisco; Ronald Petersen, MD, PhD, Principal Investigator — Mayo Clinic - Rochester, Minnesota; Paul Aisen, MD, Principal Investigator — University of California, San Diego
Locations (59):
- United States (54):
  - University of Alabama, Birmingham, Alabama
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Sun Health / Arizona Consortium, Sun City, Arizona
  - University of California, Irvine, Irvine, California
  - University of California, Irvine - Brain Imaging Center, Irvine, California
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Olin Neuropsychiatry Research Center, Hartford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Wein Center, Miami, Florida
  - Byrd Alzheimer's Institute, Tampa, Florida
  - Premiere Neurological Group, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center/Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University Schools of Medicine and Public Health, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - Dent Neurological Institute, Amherst, New York
  - New York University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - Dent Neurological Institute, Orchard Park, New York
  - University of Rochester Medical Center, Rochester, New York
  - Neurological Care of CNY, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, North Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Canada (5):
  - University of British Columbia, Vancouver, British Columbia
  - Parkwood Hospital, London, Ontario
  - Saint Joseph's Hospital, London, Ontario
  - Sunnybrook and Women's College, Health Sciences Centre, University of Toronto, Toronto, Ontario
  - Jewish Hospital Memory Clinic, Quebec, Montreal, Quebec

REFERENCES:
- [Background] Frank RA, Galasko D, Hampel H, Hardy J, de Leon MJ, Mehta PD, Rogers J, Siemers E, Trojanowski JQ; National Institute on Aging Biological Markers Working Group. Biological markers for therapeutic trials in Alzheimer's disease. Proceedings of the biological markers working group; NIA initiative on neuroimaging in Alzheimer's disease. Neurobiol Aging. 2003 Jul-Aug;24(4):521-36. doi: 10.1016/s0197-4580(03)00002-2. No abstract available. PMID 12714109
- [Background] Grundman M, Petersen RC, Ferris SH, Thomas RG, Aisen PS, Bennett DA, Foster NL, Jack CR Jr, Galasko DR, Doody R, Kaye J, Sano M, Mohs R, Gauthier S, Kim HT, Jin S, Schultz AN, Schafer K, Mulnard R, van Dyck CH, Mintzer J, Zamrini EY, Cahn-Weiner D, Thal LJ; Alzheimer's Disease Cooperative Study. Mild cognitive impairment can be distinguished from Alzheimer disease and normal aging for clinical trials. Arch Neurol. 2004 Jan;61(1):59-66. doi: 10.1001/archneur.61.1.59. PMID 14732621
- [Background] Petersen RC. Mild cognitive impairment clinical trials. Nat Rev Drug Discov. 2003 Aug;2(8):646-53. doi: 10.1038/nrd1155. No abstract available. PMID 12904814
- [Derived] Mukesha D, Firat H, Sacco G. Integrating large-scale serum metabolomics and APOE epsilon4 genotype status for the non-invasive detection of Alzheimer's disease in the ADNI cohort. medRxiv [Preprint]. 2026 Jan 16:2025.12.29.25343146. doi: 10.64898/2025.12.29.25343146. PMID 41646720
- [Derived] Gong Z, Laporte JP, Guo AY, Bilgel M, Bae J, Fox NY, de Rouen A, Zhang N, Taranath A, de Cabo R, Egan JM, Ferrucci L, Bouhrara M. Early axonal degeneration linked to clinical decline in Alzheimer's disease progression revealed with diffusion MRI. J Clin Invest. 2025 Nov 27:e196638. doi: 10.1172/JCI196638. Online ahead of print. PMID 41307953
- [Derived] Yang S, Zhang X, Du X, Yan P, Zhang J, Wang W, Wang J, Zhang L, Sun H, Liu Y, Xu X, Di Y, Zhong J, Wu C, Reinhardt JD, Zheng Y, Wu T. Prediction of cognitive conversion within the Alzheimer's disease continuum using deep learning. Alzheimers Res Ther. 2025 Feb 13;17(1):41. doi: 10.1186/s13195-025-01686-x. PMID 39948600
- [Derived] Miller AA, Sharp ES, Wang S, Zhao Y, Mecca AP, van Dyck CH, O'Dell RS; Alzheimer's Disease Neuroimaging Initiative (ADNI). Self-reported hearing loss is associated with faster cognitive and functional decline but not diagnostic conversion in the ADNI cohort. Alzheimers Dement. 2024 Nov;20(11):7847-7858. doi: 10.1002/alz.14252. Epub 2024 Sep 26. PMID 39324520
- [Derived] Cullen NC, Leuzy A, Palmqvist S, Janelidze S, Stomrud E, Pesini P, Sarasa L, Allue JA, Proctor NK, Zetterberg H, Dage JL, Blennow K, Mattsson-Carlgren N, Hansson O. Individualized prognosis of cognitive decline and dementia in mild cognitive impairment based on plasma biomarker combinations. Nat Aging. 2021 Jan;1(1):114-123. doi: 10.1038/s43587-020-00003-5. Epub 2020 Nov 30. PMID 37117993
- [Derived] Klingenberg M, Stark D, Eitel F, Budding C, Habes M, Ritter K; Alzheimer's Disease Neuroimaging Initiative. Higher performance for women than men in MRI-based Alzheimer's disease detection. Alzheimers Res Ther. 2023 Apr 20;15(1):84. doi: 10.1186/s13195-023-01225-6. PMID 37081528
- [Derived] Behzad M, Zirak N, Madani GH, Baidoo L, Rezaei A, Karbasi S, Sadeghi M, Shafie M, Mayeli M, Alzheimer's Disease Neuroimaging Initiative. CSF-Targeted Proteomics Indicate Amyloid-Beta Ratios in Patients with Alzheimer's Dementia Spectrum. Int J Alzheimers Dis. 2023 Feb 6;2023:5336273. doi: 10.1155/2023/5336273. eCollection 2023. PMID 36793451
- [Derived] Rouch L, Virecoulon Giudici K, Cantet C, Guyonnet S, Delrieu J, Legrand P, Catheline D, Andrieu S, Weiner M, de Souto Barreto P, Vellas B; Alzheimer's Disease Neuroimaging Initiative. Associations of erythrocyte omega-3 fatty acids with cognition, brain imaging and biomarkers in the Alzheimer's disease neuroimaging initiative: cross-sectional and longitudinal retrospective analyses. Am J Clin Nutr. 2022 Dec 19;116(6):1492-1506. doi: 10.1093/ajcn/nqac236. PMID 36253968
- [Derived] Xu G, Zheng S, Zhu Z, Yu X, Jiang J, Jiang J, Chu Z; Alzheimer's Disease Neuroimaging Initiative. Association of tau accumulation and atrophy in mild cognitive impairment: a longitudinal study. Ann Nucl Med. 2020 Nov;34(11):815-823. doi: 10.1007/s12149-020-01506-2. Epub 2020 Aug 12. PMID 32785820
- [Derived] Kennedy RE, Schneider LS, Cutter GR; Alzheimer's Disease Neuroimaging Initiative. Biomarker positive and negative subjects in the ADNI cohort: clinical characterization. Curr Alzheimer Res. 2012 Dec;9(10):1135-41. doi: 10.2174/156720512804142976. PMID 22963265
- [Derived] Grill JD, Di L, Lu PH, Lee C, Ringman J, Apostolova LG, Chow N, Kohannim O, Cummings JL, Thompson PM, Elashoff D; Alzheimer's Disease Neuroimaging Initiative. Estimating sample sizes for predementia Alzheimer's trials based on the Alzheimer's Disease Neuroimaging Initiative. Neurobiol Aging. 2013 Jan;34(1):62-72. doi: 10.1016/j.neurobiolaging.2012.03.006. Epub 2012 Apr 13. PMID 22503160
- [Derived] Schrag A, Schott JM; Alzheimer's Disease Neuroimaging Initiative. What is the clinically relevant change on the ADAS-Cog? J Neurol Neurosurg Psychiatry. 2012 Feb;83(2):171-3. doi: 10.1136/jnnp-2011-300881. Epub 2011 Oct 21. PMID 22019547
- [Derived] Samtani MN, Farnum M, Lobanov V, Yang E, Raghavan N, Dibernardo A, Narayan V; Alzheimer's Disease Neuroimaging Initiative. An improved model for disease progression in patients from the Alzheimer's disease neuroimaging initiative. J Clin Pharmacol. 2012 May;52(5):629-44. doi: 10.1177/0091270011405497. Epub 2011 Jun 9. PMID 21659625
- [Derived] Schneider LS, Insel PS, Weiner MW; Alzheimer's Disease Neuroimaging Initiative. Treatment with cholinesterase inhibitors and memantine of patients in the Alzheimer's Disease Neuroimaging Initiative. Arch Neurol. 2011 Jan;68(1):58-66. doi: 10.1001/archneurol.2010.343. PMID 21220675
- [Derived] Schneider LS, Kennedy RE, Cutter GR; Alzheimer's Disease Neuroimaging Initiative. Requiring an amyloid-beta1-42 biomarker for prodromal Alzheimer's disease or mild cognitive impairment does not lead to more efficient clinical trials. Alzheimers Dement. 2010 Sep;6(5):367-77. doi: 10.1016/j.jalz.2010.07.004. PMID 20813339
- See also: Alzheimer's Disease Neuroimaging Initiative--Additional Information — http://www.alzheimers.org/clintrials/ADNI.htm
- See also: Laboratory of Neuro Imaging: Alzheimer's Disease Neuroimaging Initiative — http://adni.loni.usc.edu/
- See also: Alzheimer's Disease Cooperative Study — http://www.adcs.org
- See also: ADEAR Center — http://www.alzheimers.org